CLINICAL TRIAL: NCT03445065
Title: Benefits of a Long Term Implantable Continuous Glucose Monitoring System for Adults With Diabetes - France Randomized Clinical Trial
Brief Title: A French Study to Evaluate the Usefulness of an Implantable Continuous Glucose Monitoring (CGM) Sensor to Improve Glycemic Control in Participants With Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Roche Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RD003329
Record Dates: First submitted 2018-02-02; First posted 2018-02-26 (Actual); Results first posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- Cohort 1, Enabled - Eversense XL CGM System (Experimental): Cohort 1 included patients with clinically confirmed diagnosis of Type 1 or Type 2 diabetes mellitus for ≥1 year and using insulin by multiple-daily subcutaneous injections or insulin pump and had an HbA1c >8%. All participants had the Eversense XL Glucose Sensor subcutaneously implanted into their arm of choice. Those randomized into the Enabled group were trained and allowed to use the Eversense XL system for continuous glucose monitoring (CGM). They were not allowed to use another CGM or FGM system.
  Interventions: Device: Eversense XL CGM System
- Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) (Active Comparator): Cohort 1 included patients with clinically confirmed diagnosis of Type 1 or Type 2 diabetes mellitus for ≥1 year and using insulin by multiple-daily subcutaneous injections or insulin pump and had an HbA1c >8%. All participants had the Eversense XL Glucose Sensor subcutaneously implanted into their arm of choice. Those randomized into the Control group were to continue using their usual glucose monitoring system (self-monitoring of blood glucose [SMBG] or flash glucose monitoring [FGM]), and the implanted Eversense XL CGM System remained in blinded mode.
  Interventions: Device: Eversense XL CGM System; Device: Usual SMBG or FGM device used by participants
- Cohort 2, Enabled - Eversense XL CGM System (Experimental): Cohort 2 included patients with Type 1 diabetes mellitus for ≥1 year and using insulin by multiple-daily subcutaneous injections or insulin pump and spending >1.5 hours per day with a sensor mean glucose of <70 mg/dL for at least 28 days (time in hypoglycemia). All participants had the Eversense XL Glucose Sensor subcutaneously implanted into their arm of choice. Those randomized into the Enabled group were trained and allowed to use the Eversense XL system for continuous glucose monitoring (CGM). They were not allowed to use another CGM or FGM system.
  Interventions: Device: Eversense XL CGM System
- Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM) (Active Comparator): Cohort 2 included patients with Type 1 diabetes mellitus for ≥1 year and using insulin by multiple-daily subcutaneous injections or insulin pump and spending >1.5 hours per day with a sensor mean glucose of <70 mg/dL for at least 28 days (time in hypoglycemia). All participants had the Eversense XL Glucose Sensor subcutaneously implanted into their arm of choice. Those randomized into the Control group were to continue using their usual glucose monitoring system (self-monitoring of blood glucose [SMBG] or flash glucose monitoring [FGM]), and the implanted Eversense XL CGM System remained in blinded mode.
  Interventions: Device: Eversense XL CGM System; Device: Usual SMBG or FGM device used by participants

INTERVENTIONS:
Device: Eversense XL CGM System — The Eversense XL Continuous Glucose Monitoring (CGM) System consists of an implantable sensor inserted under the skin, an external transmitter, and a Mobile Medical Application (MMA) for display of glucose information that runs on a Handheld Device (HHD).
Device: Usual SMBG or FGM device used by participants — Commercially available products in France for self-monitoring of blood glucose (SMBG) or flash glucose monitoring (FGM) were considered as comparators for this study.
  Arms: Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM); Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)

SUMMARY:
This study will be conducted in France and will evaluate the usefulness of using a long-term subcutaneously inserted continuous glucose monitoring (CGM) sensor (the Eversense XL CGM System) to improve glycemic control in patients with either Type 1 or Type 2 diabetes mellitus under insulin therapy. Participants will be enrolled into one of two cohorts (Cohorts 1 and 2). Cohort 1 will be focused on participants with Type 1 or Type 2 diabetes with hemoglobin A1C (HbA1c) >8%. Cohort 2 will be focused on participants with Type 1 diabetes spending more than 1.5 hours per day with mean glucose <70 mg/dL, including excursions below 54 mg/dL, for at least 28 days. Within each cohort, participants will be randomized in a 2:1 ratio to one of two groups: the Enabled and Control groups, respectively. The Enabled group will be trained to use the CGM system, whereas the Control group will continue with their usual glucose monitoring system (self-monitoring of blood glucose [SMBG] or flash glucose monitoring [FGM]).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants at least 18 years of age
* Clinically confirmed diagnosis of Type 1 or Type 2 diabetes mellitus for ≥1 year and using insulin by multiple-daily subcutaneous injections or insulin pump and an HbA1c > 8% (Cohort 1)
* Clinically confirmed diagnosis of Type 1 diabetes mellitus for ≥1 year and using insulin by multiple-daily subcutaneous injections or insulin pump and spending more than more than 1.5 hour with sensor glucose <70 mg/dl per day including excursions below 54 mg/dl as a mean for at least 28 days (Cohort 2)
* Participant is willing to comply with protocol

Exclusion Criteria:

* Female participants of childbearing capacity (defined as not surgically sterile or not menopausal for ≥ 1 year) who are lactating or pregnant, intending to become pregnant, or not practicing birth control during the course of the study
* A condition preventing or complicating the placement, operation or removal of the Sensor or wearing of transmitter, including upper extremity deformities or skin condition
* History of hepatitis B, hepatitis C, or HIV
* Currently receiving (or likely to need during the study period): immunosuppressant therapy; chemotherapy; anticoagulant/antithrombotic therapy (excluding aspirin < 2000 mg per day); antibiotics for chronic infection (e.g. osteomyelitis, endocarditis)
* A condition requiring or likely to require magnetic resonance imaging (MRI)
* Known topical or local anesthetic allergy
* Known allergy to glucocorticoids or using systemic glucocorticoids (excluding topical, optical or nasal but including inhaled)
* Any condition that in the investigator's opinion would make the participant unable to complete the study or would make it not in the participant's best interest to participate in the study. Conditions include, but are not limited to, psychiatric conditions, known current or recent alcohol abuse or drug abuse by participant history, a condition that may increase the risk of induced hypoglycemia or risk related to repeated blood testing. Investigator will supply rationale for exclusion
* Participation in another clinical investigation (drug or device) within 2 weeks prior to screening or intent to participate during the study period
* Legal incompetence or limited legal competence
* Dependency on sponsor or Investigator (e.g. co-worker or family member)
* The presence of any other active implanted device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Berteau, Study Director — Hoffmann-La Roche
Locations (20):
- France (20):
  - CHU Amiens Picardie, Amiens
  - CHU Caen Normandie, Caen
  - CHU Grenoble Alpes, La Tronche
  - Hopital Hotel Dieu - Creusot, Le Creusot
  - CHRU de Lille, Lille
  - APHM - Hopital Sainte-Marguerite, Marseille
  - CHU de Montpellier, Montpellier
  - Hopital Caremeau-CHU Nimes, Nîmes
  - Paris Lariboisière, Paris
  - APHP Groupe Hospitalier Cochin (Paris), Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Rouen, Rouen
  - CHU de Nantes, Saint-Herblain
  - CHRU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHU de Nancy, Vandœuvre-lès-Nancy
  - Institut de diabétologie et Nutrition du Centre, Vernouillet
  - Groupe hospitalier Les Portes du Sud, Vénissieux

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM): Cohort 2 included patients with Type 1 diabetes mellitus for ≥1 year and using insulin by multiple-daily subcutaneous injections or insulin pump and spending >1.5 hours per day with a sensor mean glucose of <70 mg/dL for at least 28 days (time in hypoglycemia). All participants had the Eversense XL Glucose Sensor subcutaneously implanted into their arm of choice. Those randomized into the Control group were to continue using their usual glucose monitoring system (self-monitoring of blood glucose [SMBG] or flash glucose monitoring [FGM]), and the implanted Eversense XL CGM System remained in blinded mode. At Day 120, participants in this Cohort 2 Control group had the opportunity to switch to have the CGM system enabled until the end of the study (Day 180).
Period: Overall Study
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Started | 97 | 52 | 62 | 28
Completed | 90 | 43 | 57 | 25
Not Completed | 7 | 9 | 5 | 3
Not completed — Withdrawal by Subject | 3 | 6 | 2 | 2
Not completed — Other | 4 | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM) | Total
Number analyzed (Participants) | 97 | 52 | 62 | 28 | 239
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (13.8) | 41.1 (13.0) | 45.1 (14.1) | 47.7 (12.7) | 44.0 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 27 | 17 | 8 | 107
  Male | 42 | 25 | 45 | 20 | 132
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Type of Diabetes [Count of Participants; unit: Participants]
  Type 1 Diabetes | 84 | 46 | 62 | 28 | 220
  Type 2 Diabetes | 13 | 6 | 0 | 0 | 19
Hemoglobin A1c (HbA1c, %) Levels at Baseline [Mean (Standard Deviation); unit: HbA1c (%)] | 9.0 (0.9) | 9.1 (0.9) | 7.3 (0.8) | 6.9 (1.0) | 8.3 (1.3)
Percentage of Time Spent in Hypoglycemia (<54 mg/dL) From Day 0 to Day 30 [Mean (Standard Deviation); unit: Percentage of time] | 1.2 (1.8) | 1.4 (2.4) | 4.7 (4.0) | 5.4 (4.5) | 2.6 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: HbA1c (%) Levels at Day 180
Description: The analysis of the primary outcome measure for Cohort 1 was an analysis of covariance (ANCOVA) comparing the HbA1c (%), defined as the percentage of hemoglobin proteins that are glycated (i.e., chemically linked to a sugar), at the Day 180 visit between the Enabled and Control arms. The statistical model included the randomization arm, center, and diabetes type as fixed classification effects, and HbA1c (%) at Day 0 as baseline covariates. Adjusted means with their 95% confidence intervals are provided.
Time Frame: Day 180
Population: This analysis of the primary outcome measure for Cohort 1 used the Full Analysis Set Population, which included all randomized participants in Cohort 1 only with sensor inserted and at least one CGM data point available. The results for Cohort 2 are presented below as a secondary outcome measure.
Measure: Mean (95% Confidence Interval); unit: HbA1c (%)
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52
HbA1c (%) | 8.6 [8.4 to 8.9] | 8.8 [8.5 to 9.0]
Statistical Analysis 1: Comparison: Cohort 1, Enabled - Eversense XL CGM System vs Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.341, ANCOVA — The significance level was set to p<0.05 (two-sided); The ANCOVA model included arm, centre, and type of diabetes as fixed classification effects, and HbA1c (%) at inclusion as baseline covariate; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.1] — The mean difference in HbA1c (%) at Day 180 was calculated as the Enabled group minus the Control group

2. Primary Outcome: Cohort 2: Percentage of Time Spent in Hypoglycemia (<54 mg/dL) From Day 90 to Day 120
Description: The analysis of the primary outcome measure for Cohort 2 was an analysis of covariance (ANCOVA) comparing the percentage of time participants in each treatment arm spent in hypoglycemia with a blood glucose level <54 milligrams per decilitre (mg/dL) between the Day 90 and Day 120 visits, based on the total duration of time with available CGM data (i.e., excluding temporary discontinuations). The statistical model included the randomization arm and center as fixed classification effects and the level of hypoglycemia at baseline (i.e. percentage of time spent in hypoglycemia <54 mg/dL between the Day 0 and Day 30 visits) as baseline covariates. Adjusted means with their 95% confidence intervals are provided.
Time Frame: From Day 90 to Day 120
Population: This analysis of the primary outcome measure for Cohort 2 used the Full Analysis Set Population, which included all randomized participants in Cohort 2 only with sensor inserted and at least one CGM data point available. The results for Cohort 1 are presented below as a secondary outcome measure.
Measure: Mean (95% Confidence Interval); unit: Percentage of time
Arm/Group | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 62 | 28
Percentage of time | 4.0 [3.0 to 5.1] | 5.7 [4.2 to 7.1]
Statistical Analysis 1: Comparison: Cohort 2, Enabled - Eversense XL CGM System vs Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.03892, ANCOVA — The significance level was set to p<0.05 (two-sided); The ANCOVA model included arm and centre as fixed classification effects and % time in hypoglycemia (<54mg/dL) Day0-30 as baseline covariate; Mean Difference (Net) = -1.6, 95% CI 2-sided [-3.1 to -0.1] — The mean difference was calculated as the Enabled group minus the Control group

3. Secondary Outcome: Number of Participants With at Least One Pre-Specified Adverse Event That Occurred Following Sensor Insertion
Time Frame: At sensor insertion (Day 0)
Population: The Safety Population included participants with sensors inserted.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Participants
  At Least One Infection, Local or Systemic | 1 | 1 | 1 | 0
  At Least One Bleeding | 0 | 0 | 0 | 1
  At Least One Edema or Swelling | 0 | 1 | 0 | 0
  At Least One Scar Formation and/or Keloid | 0 | 0 | 0 | 0
  At Least One Skin Irritation and/or Redness | 4 | 1 | 1 | 0
  At Least One Nerve Damage Causing Tingling, Numbness, Pain, or Weakness | 1 | 0 | 0 | 0
  At Least One Itching and/or Pruritus | 2 | 0 | 2 | 1
  At Least One Discoloration of Skin | 0 | 1 | 0 | 0
  At Least One Hematoma Formation | 0 | 2 | 3 | 0
  At Least One Pain and/or Burning Sensation | 1 | 1 | 0 | 0
  At Least One Device Migration | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With at Least One Pre-Specified Adverse Event That Occurred Following Sensor Removal
Time Frame: At sensor removal (up to Day 180)
Population: The Safety Population included participants with sensors inserted.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Participants
  At Least One Infection, Local or Systemic | 0 | 0 | 0 | 0
  At Least One Bleeding | 0 | 0 | 0 | 0
  At Least One Edema or Swelling | 0 | 0 | 0 | 0
  At Least One Scar Formation and/or Keloid | 0 | 0 | 0 | 0
  At Least One Skin Irritation and/or Redness | 0 | 0 | 0 | 0
  At Least One Nerve Damage Causing Tingling, Numbness, Pain, or Weakness | 0 | 0 | 0 | 0
  At Least One Itching and/or Pruritus | 0 | 0 | 0 | 0
  At Least One Discoloration of Skin | 0 | 0 | 0 | 0
  At Least One Hematoma Formation | 0 | 1 | 0 | 0
  At Least One Pain and/or Burning Sensation | 1 | 1 | 1 | 0
  At Least One Device Migration | 0 | 0 | 0 | 0

5. Secondary Outcome: Overall Number of Participants With at Least One Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in participants, whether or not related to the investigational medical device. AEs were coded using the MedDRA dictionary version 20.1. All AEs were assessed by the investigator for relation to the device, seriousness (according to serious AE criteria), and severity (i.e., intensity of the event: mild, moderate, or severe). AEs of hypoglycemia were identified using a Standardized MedDRA Query (SMQ) for a list of Preferred Terms; all terms for hypoglycemia reported in the AE forms were considered symptomatic hypoglycemia. 'Severe hypoglycemia' included all serious and severe/life-threatening events of the SMQ for hypoglycemia. Serious diabetic ketoacidosis was identified in the AE forms using a set list of MedDRA terms. Adverse device effects (ADEs) included all AEs that were pre-specified in the electronic Case Report Form (eCRF).
Time Frame: From Day 0 (Insertion) up to Day 180; for Cohort 2, Contol: From Day 0 to Day 120 and From Day 120 to Day 180
Population: The Safety Population included participants with sensors inserted.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2, Control (Day 0 to 120) - Usual Glucose Monitoring System (SMBG or FGM): Cohort 2 included patients with Type 1 diabetes mellitus for ≥1 year and using insulin by multiple-daily subcutaneous injections or insulin pump and spending >1.5 hours per day with a sensor mean glucose of <70 mg/dL for at least 28 days (time in hypoglycemia). All participants had the Eversense XL Glucose Sensor subcutaneously implanted into their arm of choice. From Day 0 to 120, those randomized into the Control group were to continue using their usual glucose monitoring system (self-monitoring of blood glucose [SMBG] or flash glucose monitoring [FGM]), and the implanted Eversense XL CGM System remained in blinded mode.
- Cohort 2, Control (Day 120 to 180) - Eversense XL CGM System or Usual Glucose Monitoring System: Cohort 2 included patients with Type 1 diabetes mellitus for ≥1 year and using insulin by multiple-daily subcutaneous injections or insulin pump and spending >1.5 hours per day with a sensor mean glucose of <70 mg/dL for at least 28 days (time in hypoglycemia). All participants had the Eversense XL Glucose Sensor subcutaneously implanted into their arm of choice. At Day 120, participants in this Cohort 2 Control group had the opportunity to switch to have the CGM system enabled until the end of the study (Day 180).
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control (Day 0 to 120) - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Control (Day 120 to 180) - Eversense XL CGM System or Usual Glucose Monitoring System
Number analyzed (Participants) | 97 | 52 | 62 | 28 | 28
Participants
  At Least One AE | 46 | 19 | 25 | 9 | 2
  At Least One Serious AE | 7 | 5 | 2 | 0 | 0
  At Least One Fatal AE | 0 | 0 | 0 | 0 | 0
  At Least One Mild AE (Maximum Severity) | 27 | 14 | 14 | 8 | 1
  At Least One Moderate AE (Maximum Severity) | 28 | 8 | 14 | 3 | 1
  At Least One Severe AE (Maximum Severity) | 6 | 5 | 2 | 0 | 0
  At Least One AE Leading to Discontinuation of Device | 2 | 4 | 0 | 1 | 0
  At Least One AE Related (Possible or Probable) to Device | 15 | 7 | 11 | 3 | 0
  At Least One AE of Symptomatic Hypoglycemia | 2 | 2 | 4 | 2 | 1
  At Least One AE of Severe Hypoglycemia | 0 | 1 | 0 | 0 | 0
  At Least One AE of Serious Diabetic Ketoacidosis | 1 | 0 | 0 | 0 | 0
  At Least One Adverse Device Effect (ADE), Collected in the eCRF | 59 | 30 | 40 | 13 | 5
  At Least One ADE, Reported to the Hotline | 39 | 17 | 28 | 7 | 5

6. Secondary Outcome: Percentage of Time Spent in the Euglycemic Range (70mg/dL-180mg/dL) From Day 90 to Day 120
Description: The results show an analysis of covariance (ANCOVA) comparing the percentage of time participants in each treatment arm of Cohorts 1 and 2 spent in euglycemia with a blood glucose level ≥70 mg/dL to ≤180 mg/dL between the Day 90 and Day 120 visits, based on the total duration of time with available CGM data (i.e., excluding temporary discontinuations). The statistical model included the randomization arm and centre (and diabetes type for Cohort 1) as fixed classification effects and the time in euglycemia at baseline (i.e. percentage of time spent in euglycemia between the Day 0 and Day 30 visits) as baseline covariates. Adjusted means with their 95% confidence intervals are provided.
Time Frame: From Day 90 to Day 120
Population: Full Analysis Set Population, which included all randomized participants with sensor inserted and at least one CGM data point available.
Measure: Mean (95% Confidence Interval); unit: Percentage of time
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Percentage of time | 47.4 [42.0 to 52.9] | 42.1 [35.8 to 48.4] | 59.8 [57.2 to 62.3] | 55.0 [51.5 to 58.6]
Statistical Analysis 1: Comparison: Cohort 1, Enabled - Eversense XL CGM System vs Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.056, ANCOVA — The significance level was set to p<0.05 (two-sided); The model included arm, centre, and diabetes type as fixed classification effects, and % time in euglycemic range (Day0-30) as baseline covariate; Mean Difference (Net) = 5.4, 95% CI 2-sided [-0.1 to 10.9] — The mean difference was calculated as the Enabled group minus the Control group
Statistical Analysis 2: Comparison: Cohort 2, Enabled - Eversense XL CGM System vs Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.01255, ANCOVA — The significance level was set to p<0.05 (two-sided); The model included arm and centre as fixed classification effects, and % time in euglycemic range (Day0-30) as baseline covariate; Mean Difference (Net) = 4.7, 95% CI 2-sided [1.0 to 8.4] — The mean difference was calculated as the Enabled group minus the Control group

7. Secondary Outcome: Percentage of Time Spent in Hyperglycemia (>250mg/dL) From Day 90 to Day 120
Description: The results show an analysis of covariance (ANCOVA) comparing the percentage of time participants in each treatment arm of Cohorts 1 and 2 spent in hyperglycemia with a blood glucose level >250 mg/dL between the Day 90 and Day 120 visits, based on the total duration of time with available CGM data (i.e., excluding temporary discontinuations). The statistical model included the randomization arm and center (and diabetes type for Cohort 1) as fixed classification effects and the level of hyperglycemia at baseline (i.e. percentage of time spent in hyperglycemia >250 mg/dL between the Day 0 and Day 30 visits) as baseline covariates. Adjusted means with their 95% confidence intervals are provided.
Time Frame: From Day 90 to Day 120
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Percentage of time
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Percentage of time | 18.5 [14.1 to 22.9] | 24.0 [19.0 to 29.1] | 8.5 [6.4 to 10.6] | 9.5 [6.7 to 12.4]
Statistical Analysis 1: Comparison: Cohort 1, Enabled - Eversense XL CGM System vs Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.015, ANCOVA — The significance level was set to p<0.05 (two-sided); Model included arm, centre, and diabetes type as fixed classification effects, and % time in hyperglycemia >250mg/dL Day0-30 as baseline covariate; Mean Difference (Net) = -5.5, 95% CI 2-sided [-9.9 to -1.1] — The mean difference was calculated as the Enabled group minus the Control group
Statistical Analysis 2: Comparison: Cohort 2, Enabled - Eversense XL CGM System vs Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.50266, ANCOVA — The significance level was set to p<0.05 (two-sided); The model included arm and centre as fixed classification effects, and % time in hyperglycemia (>250mg/dL) Day0-30 as baseline covariate; Mean Difference (Net) = -1.0, 95% CI 2-sided [-4.0 to 2.0] — The mean difference was calculated as the Enabled group minus the Control group

8. Secondary Outcome: Percentage of Time Spent in Hyperglycemia (>180mg/dL) From Day 90 to Day 120
Description: The results show an analysis of covariance (ANCOVA) comparing the percentage of time participants in each treatment arm of Cohorts 1 and 2 spent in hyperglycemia with a blood glucose level >180 mg/dL between the Day 90 and Day 120 visits, based on the total duration of time with available CGM data (i.e., excluding temporary discontinuations). The statistical model included the randomization arm and center (and diabetes type for Cohort 1) as fixed classification effects and the level of hyperglycemia at baseline (i.e. percentage of time spent in hyperglycemia >180 mg/dL between the Day 0 and Day 30 visits) as baseline covariate. Adjusted means with their 95% confidence intervals are provided.
Time Frame: From Day 90 to Day 120
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Percentage of time
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Percentage of time | 50.0 [44.3 to 55.8] | 55.2 [48.6 to 61.8] | 30.7 [28.0 to 33.5] | 34.0 [30.2 to 37.9]
Statistical Analysis 1: Comparison: Cohort 1, Enabled - Eversense XL CGM System vs Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.080, ANCOVA — The significance level was set to p<0.05 (two-sided); Model included arm, centre, and diabetes type as fixed classification effects, and % time in hyperglycemia >180mg/dL Day0-30 as baseline covariate; Mean Difference (Net) = -5.1, 95% CI 2-sided [-10.9 to 0.6] — The mean difference was calculated as the Enabled group minus the Control group
Statistical Analysis 2: Comparison: Cohort 2, Enabled - Eversense XL CGM System vs Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.10637, ANCOVA — The significance level was set to p<0.05 (two-sided); The model included arm and centre as fixed classification effects, and % time in hyperglycemia (>180mg/dL) Day0-30 as baseline covariate; Mean Difference (Net) = -3.3, 95% CI 2-sided [-7.3 to 0.7] — The mean difference was calculated as the Enabled group minus the Control group

9. Secondary Outcome: Percentage of Time Spent in Hypoglycemia (<70mg/dL) From Day 90 to Day 120
Description: The results show an analysis of covariance (ANCOVA) comparing the percentage of time participants in each treatment arm of Cohort 1 spent in hypoglycemia with a blood glucose level <70 mg/dL between the Day 90 and Day 120 visits, based on the total duration of time with available CGM data (i.e., excluding temporary discontinuations). The statistical model included the randomization arm and center (and diabetes type for Cohort 1) as fixed classification effects and the level of hypoglycemia at baseline (i.e. percentage of time spent in hypoglycemia <70 mg/dL between the Day 0 and Day 30 visits) as baseline covariate. Adjusted means with their 95% confidence intervals are provided.
Time Frame: From Day 90 to Day 120
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Percentage of time
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Percentage of time | 2.6 [1.6 to 3.5] | 2.8 [1.7 to 3.9] | 9.5 [7.9 to 11.1] | 11.3 [9.1 to 13.5]
Statistical Analysis 1: Comparison: Cohort 1, Enabled - Eversense XL CGM System vs Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.671, ANCOVA — The significance level was set to p<0.05 (two-sided); Model included arm, centre, and diabetes type as fixed classification effects, and % time in hypoglycemia (<70mg/dL) Day0-30 as baseline covariate; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.2 to 0.7] — The mean difference was calculated as the Enabled group minus the Control group
Statistical Analysis 2: Comparison: Cohort 2, Enabled - Eversense XL CGM System vs Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.12935, ANCOVA — The significance level was set to p<0.05 (two-sided); The model included arm and centre as fixed classification effects, and % time in hypoglycemia (<70mg/dL) Day0-30 as baseline covariate; Mean Difference (Net) = -1.8, 95% CI 2-sided [-4.1 to 0.5] — The mean difference was calculated as the Enabled group minus the Control group

10. Secondary Outcome: Cohort 1: Percentage of Time Spent in Hypoglycemia (<54mg/dL) From Day 90 to Day 120
Description: The results show an analysis of covariance (ANCOVA) comparing the percentage of time participants in each treatment arm of Cohort 1 spent in hypoglycemia with a blood glucose level <54 mg/dL between the Day 90 and Day 120 visits, based on the total duration of time with available CGM data (i.e., excluding temporary discontinuations). The statistical model included the randomization arm, center, and diabetes type as fixed classification effects and the level of hypoglycemia at baseline (i.e. percentage of time spent in hypoglycemia <54 mg/dL between the Day 0 and Day 30 visits) as baseline covariate. Adjusted means with their 95% confidence intervals are provided.
Time Frame: From Day 90 to Day 120
Population: The analysis of this secondary outcome measure for Cohort 1 used the Full Analysis Set Population, which included all randomized participants in Cohort 1 only with sensor inserted and at least one CGM data point available. The results for Cohort 2 are presented as a primary outcome measure.
Measure: Mean (95% Confidence Interval); unit: Percentage of time
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52
Percentage of time | 1.1 [0.5 to 1.6] | 1.2 [0.5 to 1.8]
Statistical Analysis 1: Comparison: Cohort 1, Enabled - Eversense XL CGM System vs Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.693, ANCOVA — The significance level was set to p<0.05 (two-sided); Model included arm, centre, and diabetes type as fixed classification effects, and % time in hypoglycemia (<54mg/dL) Day0-30 as baseline covariate; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.6 to 0.4] — The mean difference was calculated as the Enabled group minus the Control group

11. Secondary Outcome: Percentage of Time Spent in the Euglycemic Range (70mg/dL-180mg/dL) From Day 150 to Day 180
Description: The results show an analysis of covariance (ANCOVA) comparing the percentage of time participants in each treatment arm of Cohorts 1 and 2 spent in euglycemia with a blood glucose level ≥70 mg/dL to ≤180 mg/dL between the Day 150 and Day 180 visits, based on the total duration of time with available CGM data (i.e., excluding temporary discontinuations). The statistical model included the randomization arm and center (and diabetes type for Cohort 1) as fixed classification effects and the level of hypoglycemia at baseline (i.e. percentage of time spent in euglycemia between the Day 0 and Day 30 visits) as baseline covariate. Adjusted means with their 95% confidence intervals are provided.
Time Frame: From Day 150 to Day 180
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Percentage of time
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Percentage of time | 47.0 [41.3 to 52.8] | 48.0 [41.4 to 54.6] | 60.7 [57.8 to 63.6] | 61.1 [57.1 to 65.1]
Statistical Analysis 1: Comparison: Cohort 1, Enabled - Eversense XL CGM System vs Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.753, ANCOVA — The significance level was set to p<0.05 (two-sided); Model included arm, centre, and diabetes type as fixed classification effects, and % time in euglycemic range (Day0-30) as baseline covariate; Mean Difference (Net) = -0.9, 95% CI 2-sided [-6.7 to 4.9] — The mean difference was calculated as the Enabled group minus the Control group
Statistical Analysis 2: Comparison: Cohort 2, Enabled - Eversense XL CGM System vs Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.84307, ANCOVA — The significance level was set to p<0.05 (two-sided); The model included arm and centre as fixed classification effect, and % time in euglycemic range (Day0-30) as baseline covariate; Mean Difference (Net) = -0.4, 95% CI 2-sided [-4.6 to 3.8] — The mean difference was calculated as the Enabled group minus the Control group

12. Secondary Outcome: Percentage of Time Spent in Hyperglycemia (>250mg/dL) From Day 150 to Day 180
Description: The results show an analysis of covariance (ANCOVA) comparing the percentage of time participants in each treatment arm of Cohorts 1 and 2 spent in hyperglycemia with a blood glucose level >250 mg/dL between the Day 150 and Day 180 visits, based on the total duration of time with available CGM data (i.e., excluding temporary discontinuations). The statistical model included the randomization arm and center (and diabetes type for Cohort 1) as fixed classification effects and the level of hypoglycemia at baseline (i.e. percentage of time spent in hyperglycemia >250 mg/dL between the Day 0 and Day 30 visits) as baseline covariates. Adjusted means with their 95% confidence intervals are provided.
Time Frame: From Day 150 to Day 180
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Percentage of time
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Percentage of time | 18.5 [14.6 to 22.5] | 19.4 [14.9 to 23.9] | 8.7 [6.9 to 10.4] | 6.3 [3.9 to 8.8]
Statistical Analysis 1: Comparison: Cohort 1, Enabled - Eversense XL CGM System vs Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.653, ANCOVA — The significance level was set to p<0.05 (two-sided); Model included arm, centre, and diabetes type as fixed classification effects, and % time in hyperglycemia (>250mg/dL) Day0-30 as baseline covariate; Mean Difference (Net) = -0.9, 95% CI 2-sided [-4.8 to 3.0] — The mean difference was calculated as the Enabled group minus the Control group
Statistical Analysis 2: Comparison: Cohort 2, Enabled - Eversense XL CGM System vs Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.07261, ANCOVA — The significance level was set to p<0.05 (two-sided); [statistical method as in outcome 7, analysis 2]; Mean Difference (Net) = 2.3, 95% CI 2-sided [-0.2 to 4.8] — The mean difference was calculated as the Enabled group minus the Control group

13. Secondary Outcome: Percentage of Time Spent in Hyperglycemia (>180mg/dL) From Day 150 to Day 180
Description: The results show an analysis of covariance (ANCOVA) comparing the percentage of time participants in each treatment arm of Cohorts 1 and 2 spent in hyperglycemia with a blood glucose level >180 mg/dL between the Day 150 and Day 180 visits, based on the total duration of time with available CGM data (i.e., excluding temporary discontinuations). The statistical model included the randomization arm and center (and diabetes type for Cohort 1) as fixed classification effects and the level of hypoglycemia at baseline (i.e. percentage of time spent in hyperglycemia >180 mg/dL between the Day 0 and Day 30 visits) as baseline covariate. Adjusted means with their 95% confidence intervals are provided.
Time Frame: From Day 150 to Day 180
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Percentage of time
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Percentage of time | 50.8 [44.7 to 56.8] | 49.5 [42.5 to 56.5] | 30.9 [27.6 to 34.2] | 27.8 [23.3 to 32.3]
Statistical Analysis 1: Comparison: Cohort 1, Enabled - Eversense XL CGM System vs Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.685, ANCOVA — The significance level was set to p<0.05 (two-sided); Model included arm, centre, and diabetes type as fixed classification effects, and % time in hyperglycemia (>180mg/dL) Day0-30 as baseline covariate; Mean Difference (Net) = 1.3, 95% CI 2-sided [-4.9 to 7.4] — The mean difference was calculated as the Enabled group minus the Control group
Statistical Analysis 2: Comparison: Cohort 2, Enabled - Eversense XL CGM System vs Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.19785, ANCOVA — The significance level was set to p<0.05 (two-sided); [statistical method as in outcome 8, analysis 2]; Mean Difference (Net) = 3.1, 95% CI 2-sided [-1.6 to 7.8] — The mean difference was calculated as the Enabled group minus the Control group

14. Secondary Outcome: Percentage of Time Spent in Hypoglycemia (<70mg/dL) From Day 150 to Day 180
Description: The results show an analysis of covariance (ANCOVA) comparing the percentage of time participants in each treatment arm of Cohorts 1 and 2 spent in hypoglycemia with a blood glucose level <70 mg/dL between the Day 150 and Day 180 visits, based on the total duration of time with available CGM data (i.e., excluding temporary discontinuations). The statistical model included the randomization arm and center (and diabetes type for Cohort 1) as fixed classification effects and the level of hypoglycemia at baseline (i.e. percentage of time spent in hypoglycemia <70 mg/dL between the Day 0 and Day 30 visits) as baseline covariate. Adjusted means with their 95% confidence intervals are provided.
Time Frame: From Day 150 to Day 180
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Percentage of time
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Percentage of time | 2.1 [0.9 to 3.2] | 2.4 [1.1 to 3.8] | 8.4 [6.3 to 10.5] | 11.7 [8.8 to 14.5]
Statistical Analysis 1: Comparison: Cohort 1, Enabled - Eversense XL CGM System vs Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.549, ANCOVA — The significance level was set to p<0.05 (two-sided); [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.5 to 0.8] — The mean difference was calculated as the Enabled group minus the Control group
Statistical Analysis 2: Comparison: Cohort 2, Enabled - Eversense XL CGM System vs Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.03180, ANCOVA — The significance level was set to p<0.05 (two-sided); [statistical method as in outcome 9, analysis 2]; Mean Difference (Net) = -3.3, 95% CI 2-sided [-6.3 to -0.3] — The mean difference was calculated as the Enabled group minus the Control group

15. Secondary Outcome: Percentage of Time Spent in Hypoglycemia (<54mg/dL) From Day 150 to Day 180
Description: The results show an analysis of covariance (ANCOVA) comparing the percentage of time participants in each treatment arm of Cohorts 1 and 2 spent in hypoglycemia with a blood glucose level <54 mg/dL between the Day 150 and Day 180 visits, based on the total duration of time with available CGM data (i.e., excluding temporary discontinuations). The statistical model included the randomization arm and center (and diabetes type for Cohort 1) as fixed classification effects and the level of hypoglycemia at baseline (i.e. percentage of time spent in hypoglycemia <54 mg/dL between the Day 0 and Day 30 visits) as baseline covariate. Adjusted means with their 95% confidence intervals are provided.
Time Frame: From Day 150 to Day 180
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Percentage of time
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Percentage of time | 1.1 [0.4 to 1.7] | 1.0 [0.3 to 1.8] | 3.4 [2.1 to 4.8] | 6.0 [4.1 to 7.9]
Statistical Analysis 1: Comparison: Cohort 1, Enabled - Eversense XL CGM System vs Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.859, ANCOVA — The significance level was set to p<0.05 (two-sided); [statistical method as in outcome 10, analysis 1]; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.6 to 0.7] — The mean difference was calculated as the Enabled group minus the Control group
Statistical Analysis 2: Comparison: Cohort 2, Enabled - Eversense XL CGM System vs Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.01124, ANCOVA — The significance level was set to p<0.05 (two-sided); The model included arm and centre as fixed classification effects, and % time in hypoglycemia (<54mg/dL) Day0-30 as baseline covariate; Mean Difference (Net) = -2.6, 95% CI 2-sided [-4.5 to -0.6] — The mean difference was calculated as the Enabled group minus the Control group

16. Secondary Outcome: Cohort 2, Enabled Arm: Percentage of Time Spent in Hypoglycemia (<54 mg/dL) During the Day 90-120 Period Compared With the Day 150-180 Period for the Enabled Group
Description: The results show an analysis of covariance (ANCOVA) comparing the percentage of time participants in the Enabled arm of Cohort 2 spent in hypoglycemia with a blood glucose level <54 mg/dL over two different time periods (between the Days 90-120 and Days 150-180), based on the total duration of time with available CGM data (i.e., excluding temporary discontinuations). The statistical model included the time period and center as fixed classification effects and the level of hypoglycemia at baseline (i.e. percentage of time spent in hypoglycemia <54 mg/dL between the Day 0 and Day 30 visits) as baseline covariate. Adjusted means with their 95% confidence intervals are provided.
Time Frame: Day 90 to Day 120; Day 150 to Day 180
Population: The analysis included all randomized participants in the Cohort 2, Enabled arm only, with sensor inserted and at least one CGM data point available.
Measure: Mean (95% Confidence Interval); unit: Percentage of time
Groups:
- Cohort 2, Enabled (Day 90 to 120) - Eversense XL CGM System; Cohort 2, Enabled (Day 150 to 180) - Eversense XL CGM System: Cohort 2 included patients with Type 1 diabetes mellitus for ≥1 year and using insulin by multiple-daily subcutaneous injections or insulin pump and spending >1.5 hours per day with a sensor mean glucose of <70 mg/dL for at least 28 days (time in hypoglycemia). All participants had the Eversense XL Glucose Sensor subcutaneously implanted into their arm of choice. Those randomized into the Enabled group were trained and allowed to use the Eversense XL system for continuous glucose monitoring (CGM). They were not allowed to use another CGM or FGM system.
Arm/Group | Cohort 2, Enabled (Day 90 to 120) - Eversense XL CGM System | Cohort 2, Enabled (Day 150 to 180) - Eversense XL CGM System
Number analyzed (Participants) | 62 | 62
Percentage of time | 4.232 [3.242 to 5.222] | 3.430 [2.469 to 4.391]
Statistical Analysis 1: Comparison: Cohort 2, Enabled (Day 90 to 120) - Eversense XL CGM System vs Cohort 2, Enabled (Day 150 to 180) - Eversense XL CGM System; Test type: Superiority; p = 0.045, Mixed Models Analysis — The significance level was set to p<0.05 (two-sided); The model included time and centre as fixed classification effects and % time in hypoglycemia (<54mg/dL) Day0-30 as baseline covariate; Mean Difference (Net) = -0.802, 95% CI 2-sided [-1.1585 to -0.018], Standard Error of Mean 0.391 — The mean difference was calculated as the Enabled (D150-180) group minus the Enabled (D90-120) group

17. Secondary Outcome: Cohort 2, Control Arm: Percentage of Time Spent in Hypoglycemia (<54 mg/dL) During the Control Period (Days 90-120) Compared With the Enabled Period (Days 150-180) for Participants Who Switched to Use the CGM System
Description: The results show an analysis of covariance (ANCOVA) comparing the percentage of time participants in the Cohort 2, Control arm spent in hypoglycemia with a blood glucose level <54 mg/dL with a different intervention over each of the two time periods (the control period, using their usual glucose monitoring system: Days 90-120, and the enabled period, using the Eversense XL CGM system: Days 150-180), based on the total duration of time with available CGM data (i.e., excluding temporary discontinuations). The statistical model included the time period and center as fixed classification effects and the level of hypoglycemia at baseline (i.e. percentage of time spent in hypoglycemia <54 mg/dL between the Day 0 and Day 30 visits) as baseline covariate. Adjusted means with their 95% confidence intervals are provided.
Time Frame: For Cohort 2, Control arm: Day 90 to Day 120; For Cohort 2, Switch from Control to Enabled arm: Day 150 to Day 180
Population: Of the Cohort 2, Control arm participants with sensor inserted and at least one CGM data point available, only the 24 participants who switched from their usual glucose monitoring system (Days 90 to 120) to use the enabled Eversense XL CGM system (Days 150 to 180) were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: Percentage of time
Groups:
- Cohort 2, Control (Day 90 to 120) - Usual Glucose Monitoring System (SMBG or FGM): Cohort 2 included patients with Type 1 diabetes mellitus for ≥1 year and using insulin by multiple-daily subcutaneous injections or insulin pump and spending >1.5 hours per day with a sensor mean glucose of <70 mg/dL for at least 28 days (time in hypoglycemia). All participants had the Eversense XL Glucose Sensor subcutaneously implanted into their arm of choice. Those randomized into the Control group were to continue using their usual glucose monitoring system (self-monitoring of blood glucose [SMBG] or flash glucose monitoring [FGM]), and the implanted Eversense XL CGM System remained in blinded mode.
- Cohort 2, Switch From Control to Enabled (Day 150 to 180) - Eversense XL CGM System: Cohort 2 included patients with Type 1 diabetes mellitus for ≥1 year and using insulin by multiple-daily subcutaneous injections or insulin pump and spending >1.5 hours per day with a sensor mean glucose of <70 mg/dL for at least 28 days (time in hypoglycemia). All participants had the Eversense XL Glucose Sensor subcutaneously implanted into their arm of choice. At Day 120, participants in this Cohort 2 Control group switched to have the CGM system enabled until the end of the study (Day 180).
Arm/Group | Cohort 2, Control (Day 90 to 120) - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Switch From Control to Enabled (Day 150 to 180) - Eversense XL CGM System
Number analyzed (Participants) | 24 | 24
Percentage of time | 5.792 [3.672 to 7.913] | 6.263 [2.737 to 9.788]
Statistical Analysis 1: Comparison: Cohort 2, Control (Day 90 to 120) - Usual Glucose Monitoring System (SMBG or FGM) vs Cohort 2, Switch From Control to Enabled (Day 150 to 180) - Eversense XL CGM System; Test type: Superiority; p = 0.763, Mixed Model for Repeated Measures — The significance level was set to p<0.05 (two-sided); [statistical method as in outcome 16, analysis 1]; Mean Difference (Net) = 0.470, 95% CI 2-sided [-2.741 to 3.682], Standard Error of Mean 1.540 — The mean difference was calculated as the Switch to Enabled (D150-180) group minus the Control (D90-120) group

18. Secondary Outcome: Glucose Variability From Day 90 to Day 120, as Estimated With a Coefficient of Variation
Description: Glucose variability was estimated with a unitless coefficient of variation, expressed as a percentage, which was computed using CGM data with the following formula: the sum of the ratios of standard deviation of daily glycemia to the mean of daily glycemia divided by the number of days with available data for the period of interest (Days 90 to 120). According to Monnier et al. Diabetes Care 2017, a coefficient of variation threshold set to 36% allows to distinguish between stable and unstable glycemia.
Time Frame: From Day 90 to Day 120
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Coefficient of variation (%)
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Coefficient of variation (%) | 29.3 [27.5 to 31.1] | 28.0 [26.0 to 30.0] | 35.8 [34.3 to 37.3] | 36.3 [34.3 to 38.3]
Statistical Analysis 1: Comparison: Cohort 1, Enabled - Eversense XL CGM System vs Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.140, ANCOVA — The significance level was set to p<0.05 (two-sided); Model included arm, centre, and diabetes type as fixed classification effects, and glucose variability Day0-30 as baseline covariate; Mean Difference (Net) = 1.3, 95% CI 2-sided [-0.4 to 3.0] — The mean difference was calculated as the Enabled group minus the Control group
Statistical Analysis 2: Comparison: Cohort 2, Enabled - Eversense XL CGM System vs Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.64110, ANCOVA — The significance level was set to p<0.05 (two-sided); The model included arm and centre as fixed classification effects, and glucose variability Day0-30 as baseline covariate; Mean Difference (Net) = -0.5, 95% CI 2-sided [-2.6 to 1.6] — The mean difference was calculated as the Enabled group minus the Control group

19. Secondary Outcome: Glucose Variability From Day 150 to Day 180, as Estimated by a Coefficient of Variation
Description: Glucose variability was estimated with a unitless coefficient of variation, expressed as a percentage, which was computed using CGM data with the following formula: the sum of the ratios of standard deviation of daily glycemia to the mean of daily glycemia divided by the number of days with available data for the period of interest (Days 150 to 180). According to Monnier et al. Diabetes Care 2017, a coefficient of variation threshold set to 36% allows to distinguish between stable and unstable glycemia.
Time Frame: From Day 150 to Day 180
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Coefficient of variation (%)
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Coefficient of variation (%) | 26.0 [23.9 to 28.1] | 25.0 [22.6 to 27.5] | 34.4 [32.8 to 36.0] | 35.1 [32.8 to 37.3]
Statistical Analysis 1: Comparison: Cohort 1, Enabled - Eversense XL CGM System vs Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.339, ANCOVA — The significance level was set to p<0.05 (two-sided); [statistical method as in outcome 18, analysis 1]; Mean Difference (Net) = 1.0, 95% CI 2-sided [-1.1 to 3.1] — The mean difference was calculated as the Enabled group minus the Control group
Statistical Analysis 2: Comparison: Cohort 2, Enabled - Eversense XL CGM System vs Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.57677, ANCOVA — The significance level was set to p<0.05 (two-sided); [statistical method as in outcome 18, analysis 2]; Mean Difference (Net) = -0.7, 95% CI 2-sided [-3.0 to 1.7] — The mean difference was calculated as the Enabled group minus the Control group

20. Secondary Outcome: HbA1c (%) Levels at Day 120
Description: The results show an analysis of covariance (ANCOVA) comparing the HbA1c (%), defined as the percentage of hemoglobin proteins that are glycated (i.e., chemically linked to a sugar), at the Day 120 visit between the Enabled and Control arms for Cohorts 1 and 2. The statistical model included the randomization arm and center (and diabetes type for Cohort 1) as fixed classification effects, and HbA1c (%) at Day 0 as baseline covariates. Adjusted means with their 95% confidence interval are provided.
Time Frame: Day 120
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: HbA1c (%)
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
HbA1c (%) | 8.6 [8.4 to 8.9] | 8.7 [8.4 to 9.0] | 7.2 [7.0 to 7.3] | 7.3 [7.0 to 7.5]
Statistical Analysis 1: Comparison: Cohort 1, Enabled - Eversense XL CGM System vs Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.558, ANCOVA — The significance level was set to p<0.05 (two-sided); The model included arm, centre, and diabetes type as fixed classification effects, and HbA1c (%) at inclusion as baseline covariate; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.3 to 0.2] — The mean difference was calculated as the Enabled group minus the Control group
Statistical Analysis 2: Comparison: Cohort 2, Enabled - Eversense XL CGM System vs Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.408, ANCOVA — The significance level was set to p<0.05 (two-sided); The model included arm and centre as fixed classification effects, and HbA1c (%) at inclusion as baseline covariate; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.3 to 0.1] — The mean difference was calculated as the Enabled group minus the Control group

21. Secondary Outcome: Cohort 2: HbA1c (%) Levels at Day 180
Description: The analysis of this secondary outcome measure for Cohort 2 was an analysis of covariance (ANCOVA) comparing the HbA1c (%), defined as the percentage of hemoglobin proteins that are glycated (i.e., chemically linked to a sugar), at the Day 180 visit between the Enabled and Control arms. The statistical model included the randomization arm and center as fixed classification effects, and HbA1c (%) at Day 0 as baseline covariates. Adjusted means with their 95% confidence interval are provided.
Time Frame: Day 180
Population: This analysis of this secondary outcome measure for Cohort 2 used the Full Analysis Set Population, which included all randomized participants in Cohort 2 only with sensor inserted and at least one CGM data point available. The results for Cohort 1 are presented as a primary outcome measure.
Measure: Mean (95% Confidence Interval); unit: HbA1c (%)
Arm/Group | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 62 | 28
HbA1c (%) | 7.2 [7.0 to 7.4] | 7.2 [6.9 to 7.4]
Statistical Analysis 1: Comparison: Cohort 2, Enabled - Eversense XL CGM System vs Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM); Test type: Superiority; p = 0.616, ANCOVA — The significance level was set to p<0.05 (two-sided); The model included arm and centre as fixed classification effects, and HbA1c (%) at inclusion as baseline covariate; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.2 to 0.4] — The mean difference in HbA1c (%) at Day 180 was calculated as the Enabled group minus the Control group

22. Secondary Outcome: Number of Participants With the First Sensor Operating at Day 150 and Day 180
Description: This measure assesses sensor life by counting the number of participants with their first inserted CGM sensor still operating at 150 days and at 180 days post-insertion. The assessment was based on the lifespan of the first sensor: for example, if lifespan of the first sensor was ≥150 days and ≥180 days, then the participant was counted as having their first sensor operating at 150 days and 180 days, respectively. The lifespan of the first inserted CGM sensor for each participant, measured in days, was calculated as the date of the last glucose measurement by the sensor minus the date of the first glucose measurement by the sensor (+1 day).
Time Frame: From Day 0 up to Day 150 and Day 180
Population: Only participants with non-missing sensor data were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Participants
  Day 150: number analyzed (Participants) | 96 | 52 | 61 | 28
  Day 150 | 73 | 27 | 40 | 19
  Day 180: number analyzed (Participants) | 96 | 52 | 61 | 28
  Day 180 | 38 | 10 | 27 | 12

23. Secondary Outcome: Mean Lifespan of the First Sensor
Description: The lifespan of the first inserted CGM sensor for each participant, measured in days, was calculated as the date of the last glucose measurement by the sensor minus the date of the first glucose measurement by the sensor (+1 day).
Time Frame: From Day 0 up to Day 180
Population: Only participants with non-missing sensor data were included in this analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 96 | 52 | 61 | 28
Days | 159.2 (33.0) | 139.8 (46.3) | 147.3 (47.8) | 156.9 (33.2)

24. Secondary Outcome: Median Number of Sensors Used by Each Participant During the Study
Time Frame: From Day 0 to Day 180
Measure: Median (Full Range); unit: Sensors per participant
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Sensors per participant | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]

25. Secondary Outcome: Number of Participants With the First Transmitter Operating at Day 150 and Day 180
Description: This measure assesses transmitter wear time by counting the number of participants with their first CGM transmitter still operating at 150 days and at 180 days after first use. The assessment was based on the lifespan of the first transmitter: for example, if lifespan of the first transmitter was ≥150 days and ≥180 days, then the participant was counted as having their first transmitter operating at 150 days and 180 days, respectively. The lifespan of the first CGM transmitter for each participant, measured in days, was calculated as the date of the last glucose measurement with the transmitter minus the date of the first glucose measurement with the transmitter (+1 day).
Time Frame: From Day 0 up to Day 150 and Day 180
Population: Only participants with non-missing transmitter data were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Participants
  Day 150: number analyzed (Participants) | 94 | 50 | 61 | 28
  Day 150 | 1 | 23 | 0 | 3
  Day 180: number analyzed (Participants) | 94 | 50 | 61 | 28
  Day 180 | 1 | 13 | 0 | 3

26. Secondary Outcome: Mean Lifespan of the First Transmitter
Description: The lifespan of the first CGM transmitter for each participant, measured in days, was calculated as the date of the last glucose measurement with the transmitter minus the date of the first glucose measurement with the transmitter (+1 day).
Time Frame: From Day 0 up to Day 180
Population: Only participants with non-missing transmitter data were included in this analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 94 | 50 | 61 | 28
Days | 34.6 (19.2) | 140.6 (46.5) | 33.8 (12.4) | 114.6 (39.2)

27. Secondary Outcome: Median Number of Transmitters Used by Each Participant During the Study
Time Frame: From Day 0 to Day 180
Measure: Median (Full Range); unit: Transmitters per participant
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Transmitters per participant | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]

28. Secondary Outcome: Number of Participants Who Accessed CGM Application Pages at Days 60, 120, and 180
Description: This was a descriptive analysis of the number of participants in the Eversense XL CGM System Enabled groups who accessed the various CGM application (app) pages/functions at study Days 60, 120, and 180. The data were collected in the electronic Case Report Form.
Time Frame: At Days 60, 120, and 180
Population: Only participants from the Enabled groups with non-missing assessments at Days 60, 120, and 180 were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 2, Enabled - Eversense XL CGM System
Number analyzed (Participants) | 97 | 62
Participants
  Day 60 - Participant uses the 'Report' function: number analyzed (Participants) | 96 | 61
  Day 60 - Participant uses the 'Report' function | 67 | 43
  Day 60 - Participant uses the 'Historic of Alerts' function: number analyzed (Participants) | 96 | 61
  Day 60 - Participant uses the 'Historic of Alerts' function | 75 | 44
  Day 60 - Participant uses the 'Log Event' function: number analyzed (Participants) | 96 | 61
  Day 60 - Participant uses the 'Log Event' function | 61 | 38
  Day 60 - Participant uses phone to look at their glucose levels: number analyzed (Participants) | 96 | 61
  Day 60 - Participant uses phone to look at their glucose levels | 95 | 61
  Day 120 - Participant uses the 'Report' function: number analyzed (Participants) | 93 | 60
  Day 120 - Participant uses the 'Report' function | 66 | 50
  Day 120 - Participant uses the 'Historic of Alerts' function: number analyzed (Participants) | 93 | 60
  Day 120 - Participant uses the 'Historic of Alerts' function | 74 | 40
  Day 120 - Participant uses the 'Log Event' function: number analyzed (Participants) | 93 | 60
  Day 120 - Participant uses the 'Log Event' function | 63 | 28
  Day 120 - Participant uses phone to look at their glucose levels: number analyzed (Participants) | 93 | 60
  Day 120 - Participant uses phone to look at their glucose levels | 89 | 58
  Day 180 - Participant uses the 'Report' function: number analyzed (Participants) | 90 | 58
  Day 180 - Participant uses the 'Report' function | 58 | 49
  Day 180 - Participant uses the 'Historic of Alerts' function: number analyzed (Participants) | 90 | 58
  Day 180 - Participant uses the 'Historic of Alerts' function | 61 | 46
  Day 180 - Participant uses the 'Log Event' function: number analyzed (Participants) | 90 | 58
  Day 180 - Participant uses the 'Log Event' function | 54 | 35
  Day 180 - Participant uses phone to look at their glucose levels: number analyzed (Participants) | 90 | 58
  Day 180 - Participant uses phone to look at their glucose levels | 81 | 55

29. Secondary Outcome: Number of Participants Issued at Least One Type of Alarm or Alert by the CGM System During the Study
Description: This outcome measure is a descriptive analysis of the number of participants who were issued various types of alarms and alerts by the Eversense XL CGM System through the mobile medical application. The alarms listed in the results table are a higher level classification for the different types of alerts that immediately follow it, until the next type of alarm is listed (for example, the 'Calibration' alarm included both 'Calibrate Now' and 'Calibration Past Due' alerts). Only participants in the Enabled groups of both cohorts actually received these alarms/alerts because the CGM remained in blinded mode for participants in the Control groups.
Time Frame: From Day 0 up to Day 180
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Participants
  At Least 1 Alarm of Any Type | 97 | 52 | 62 | 28
  At Least 1 'Calibration' Alarm | 97 | 52 | 62 | 28
  At Least 1 'Calibrate Now' Alert | 97 | 52 | 62 | 28
  At Least 1 'Calibration Past Due' Alert | 95 | 50 | 61 | 26
  At Least 1 'Sensor Glucose' Alarm | 95 | 2 | 61 | 22
  At Least 1 'High Glucose' Alert | 95 | 2 | 61 | 22
  At Least 1 'Low Glucose' Alert | 94 | 2 | 61 | 22
  At Least 1 'Out of Range High Glucose' Alert | 86 | 1 | 47 | 8
  At Least 1 'Out of Range Low Glucose' Alert | 84 | 2 | 61 | 22
  At Least 1 'Predicted High Glucose' Alert | 44 | 1 | 39 | 8
  At Least 1 'Predicted Low Glucose' Alert | 44 | 1 | 38 | 8
  At Least 1 'Rate Falling' Alert | 31 | 1 | 27 | 6
  At Least 1 'Rate Rising' Alert | 31 | 1 | 27 | 6
  At Least 1 'Sensor Glucose and Calibration' Alarm | 31 | 19 | 18 | 10
  At Least 1 'Sensor Check' Alert | 31 | 19 | 18 | 10
  At Least 1 'Sensor Related' Alarm | 97 | 52 | 62 | 28
  At Least 1 'High Ambient Light Alert' Alert | 84 | 40 | 47 | 19
  At Least 1 'High Sensor Temperature' Alert | 1 | 1 | 3 | 0
  At Least 1 'Low Sensor Temperature' Alert | 7 | 4 | 4 | 4
  At Least 1 'New Sensor Detected' Alert | 95 | 51 | 62 | 28
  At Least 1 'Sensor Replacement' Alert | 93 | 46 | 58 | 27
  At Least 1 'System Related' Alarm, 'Displayed on the Status Bar of the App' Alert | 97 | 52 | 62 | 28
  At Least 1 'Transmitter Related' Alarm | 97 | 52 | 62 | 28
  At Least 1 'Battery Empty' Alert | 82 | 44 | 57 | 21
  At Least 1 'Charge Transmitter' Alert | 94 | 49 | 59 | 28
  At Least 1 'High Transmitter Temperature' Alert | 21 | 11 | 16 | 4
  At Least 1 'Transmitter Disconnect' Alert | 97 | 52 | 62 | 28
  At Least 1 'Transmitter Error' Alert | 9 | 2 | 6 | 3

30. Secondary Outcome: Diabetes Treatment Satisfaction Questionnaire - Original Status (DTSQs) Treatment Satisfaction Score at Baseline, Day 60, and Day 180
Description: The DTSQs questionnaire contains eight items scored on a 7-point scale (i.e. each item is scored from 0 to 6). Six items measure Treatment Satisfaction, dealing with: satisfaction with current treatment; convenience of the treatment; flexibility; satisfaction with own understanding of participant's diabetes; how likely to recommend their present treatment; and how satisfied to continue with their present treatment. These are summed to produce a total Treatment Satisfaction score, with a minimum value of 0 and a maximum value of 36; a higher score indicates greater treatment satisfaction. In case of missing items, the overall score was calculated as the mean of the available items.
Time Frame: Baseline (Day 0), Day 60, and Day 180
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Score on a scale
  Baseline | 27.0 (6.0) | 24.4 (6.3) | 26.4 (5.4) | 26.8 (5.7)
  Day 60 | 28.3 (5.8) | 24.3 (5.9) | 27.9 (4.9) | 24.4 (6.1)
  Day 180 | 26.8 (6.4) | 24.5 (7.1) | 27.6 (4.2) | 26.2 (6.1)

31. Secondary Outcome: Change From Baseline in the DTSQs Treatment Satisfaction Score at Day 60 and Day 180
Description: The DTSQs questionnaire contains eight items scored on a 7-point scale (i.e. each item is scored from 0 to 6). Six items measure Treatment Satisfaction (dealing with: satisfaction with current treatment; convenience of the treatment; flexibility; satisfaction with own understanding of participant's diabetes; how likely to recommend their present treatment; and how satisfied to continue with their present treatment). These are summed to produce a total Treatment Satisfaction score, with a minimum value of 0 and a maximum value of 36; a higher score indicates greater treatment satisfaction. For the change from baseline analysis, a positive value indicates an improvement in treatment satisfaction. In case of missing items, the overall score was calculated as the mean of the available items.
Time Frame: Baseline (Day 0), Day 60, and Day 180
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Score on a scale
  Change from Baseline at Day 60 | 1.3 (5.1) | 0.2 (6.3) | 1.7 (5.5) | -1.8 (4.1)
  Change from Baseline at Day 180 | -0.1 (6.4) | -0.1 (6.6) | 1.3 (4.4) | -0.1 (4.8)

32. Secondary Outcome: Diabetes Treatment Satisfaction Questionnaire - Change Version (DTSQc) Treatment Satisfaction Score at Day 180
Description: The DTSQc questionnaire contains eight items scored on a 7-point scale (i.e. each item is scored from -3 to +3). Six items measure Treatment Satisfaction (dealing with: satisfaction with current treatment; convenience of the treatment; flexibility; satisfaction with own understanding of participant's diabetes; how likely to recommend their present treatment; and how satisfied to continue with their present treatment). These are summed to produce a total Treatment Satisfaction score, with a minimum value of -18 and a maximum value of +18; a higher score indicates greater treatment satisfaction. In case of missing items, the overall score was calculated as the mean of the available items.
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Score on a scale | 8.6 (7.8) | 7.1 (7.0) | 8.6 (6.6) | 5.3 (8.7)

33. Secondary Outcome: Audit of Diabetes-Dependent Quality of Life (ADDQoL) Score at Baseline and Day 180
Description: The ADDQoL measures the impact of diabetes and its treatment on 19 specific aspects of life. The scale ranges from -3 to +1 for 19 life domains (impact rating) and from 0 to +3 in attributed importance (importance rating). A weighted score for each domain is calculated as a multiplier of impact rating and importance rating (ranging from -9 to +3). Finally, a mean weighted impact score (ADDQOL score) is calculated for the entire scale across all applicable domains; a higher score indicates greater quality of life.
Time Frame: Baseline (Day 0) and Day 180
Population: Only participants with non-missing data at each timepoint were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Score on a scale
  Baseline: number analyzed (Participants) | 89 | 50 | 58 | 25
  Baseline | -2.9 (1.9) | -3.0 (1.6) | -2.7 (1.9) | -1.9 (1.4)
  Day 180: number analyzed (Participants) | 65 | 33 | 45 | 22
  Day 180 | -2.7 (1.9) | -3.2 (2.1) | -2.5 (1.7) | -1.4 (1.2)

34. Secondary Outcome: Change From Baseline in the Audit of Diabetes-Dependent Quality of Life (ADDQoL) Score at Day 180
Description: The ADDQoL measures the impact of diabetes and its treatment on 19 specific aspects of life. The scale ranges from -3 to +1 for 19 life domains (impact rating) and from 0 to +3 in attributed importance (importance rating). A weighted score for each domain is calculated as a multiplier of impact rating and importance rating (ranging from -9 to +3). Finally, a mean weighted impact score (ADDQOL score) is calculated for the entire scale across all applicable domains; a higher score indicates greater quality of life. For the change from baseline analysis, a positive value indicates an improvement in quality of life.
Time Frame: Baseline (Day 0) and Day 180
Population: Only participants with non-missing data at Baseline and Day 180 were included in this analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 64 | 33 | 45 | 21
Score on a scale | 0.1 (1.4) | 0.0 (1.0) | 0.1 (1.1) | 0.4 (1.2)

35. Secondary Outcome: The Continuous Glucose Monitoring Satisfaction (CGM-SAT) Questionnaire Overall Score at Day 60 and Day 180
Description: The CGM-SAT questionnaire comprises 44 item scales assessing experiences with CGM over the previous 6 months. The scale is designed to measure the impact of CGM on diabetes management and family relationships, plus on satisfaction with emotional, behavioral and cognitive effects of CGM use. The responses were rated on a 5-point scale from '1 = strongly agree' to '5 = strongly disagree'. The overall score corresponds to the mean of the 44 items of potential positive or negative effects of using the CGM device; a higher score reflects more favorable impact of, and satisfaction with CGM. In case of missing items, the overall score was calculated as the mean of the available items.
Time Frame: Day 60 and Day 180
Population: The CGM-SAT questionnaire was completed only by participants in the Enabled groups in Cohorts 1 and 2. Only participants who completed at least one item at Day 60 or Day 180 were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 2, Enabled - Eversense XL CGM System
Number analyzed (Participants) | 97 | 62
Score on a scale
  Day 60: number analyzed (Participants) | 85 | 52
  Day 60 | 2.9 (0.3) | 3.0 (0.3)
  Day 180: number analyzed (Participants) | 63 | 44
  Day 180 | 2.8 (0.3) | 2.8 (0.3)

36. Secondary Outcome: Change From Day 60 in the CGM-SAT Questionnaire Overall Score at Day 180
Description: The CGM-SAT questionnaire comprises 44 item scales assessing experiences with CGM over the previous 6 months. The scale is designed to measure the impact of CGM on diabetes management and family relationships, plus on satisfaction with emotional, behavioral and cognitive effects of CGM use. The responses were rated on a 5-point scale from '1 = strongly agree' to '5 = strongly disagree'. The overall score corresponds to the mean of the 44 items of potential positive or negative effects of using the CGM device; a higher score (or positive change from baseline score) reflects more favorable impact of, and satisfaction with CGM. In case of missing items, the overall score was calculated as the mean of the available items.
Time Frame: Day 60 and Day 180
Population: The CGM-SAT questionnaire was completed only by participants in the Enabled groups in Cohorts 1 and 2. Only participants who completed at least one item at both Days 60 and 180 were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 2, Enabled - Eversense XL CGM System
Number analyzed (Participants) | 62 | 42
Score on a scale | -0.1 (0.3) | -0.1 (0.2)

37. Secondary Outcome: Diabetes Distress Scale 2 (DDS2) Questionnaire Score at Baseline, Day 60, and Day 180
Description: The DDS2 is a 2-item diabetes distress screening instrument asking respondents to rate on a 6-point scale (from 1 = 'Not a problem' to 6 = 'A very serious problem') the degree to which the following items caused distress: (1) feeling overwhelmed by the demands of living with diabetes, and (2) feeling that I am often failing with my diabetes regimen. The DDS2 score is the mean of the two items (ranging from 1 to 6). A lower DDS2 score (or a negative change from baseline score) indicates a lower level of distress. If one item was missing, then no score was computed.
Time Frame: Baseline (Day 0), Day 60, and Day 180
Population: Only participants with non-missing data at each timepoint were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Score on a scale
  Baseline: number analyzed (Participants) | 22 | 13 | 16 | 7
  Baseline | 2.4 (1.1) | 3.1 (1.6) | 2.8 (1.2) | 2.3 (1.0)
  Day 60: number analyzed (Participants) | 21 | 13 | 14 | 5
  Day 60 | 2.1 (1.0) | 3.0 (1.2) | 2.6 (1.5) | 3.0 (2.0)
  Day 180: number analyzed (Participants) | 17 | 8 | 14 | 6
  Day 180 | 2.1 (1.2) | 2.6 (1.1) | 2.4 (1.3) | 2.0 (1.1)

38. Secondary Outcome: Change From Baseline in the Diabetes Distress Scale 2 (DDS2) Questionnaire Score at Day 60 and Day 180
Description: as for outcome 37
Time Frame: Baseline (Day 0), Day 60, and Day 180
Population: Only participants with non-missing data at Baseline and Day 60 or Day 180 were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 21 | 13 | 14 | 5
Score on a scale
  Change from Baseline at Day 60 | -0.2 (0.8) | 0.0 (1.2) | -0.3 (2.1) | 0.6 (1.4)
  Change from Baseline at Day 180: number analyzed (Participants) | 17 | 8 | 14 | 5
  Change from Baseline at Day 180 | -0.2 (0.9) | -0.6 (1.5) | -0.5 (1.9) | 0.0 (0.8)

39. Secondary Outcome: Hypoglycemia Fear Survey, Part 2 (HFS2) Worry Subscale Score at Baseline, Day 60, and Day 180
Description: HFS2 Worry items describe specific concerns that patients may have about their hypoglycemic episodes (e.g., being alone, episodes occurring during sleep, or having an accident). The 5-point Likert scale for each item ranges from 0 (never) to 4 (almost always), and the HFS2 Worry subscale score is the sum of all 18 items (ranging from 0 to 72). A lower HFS2 Worry subscale score (or a negative change from baseline score) indicates a lower level of fear of hypoglycemia. There was no plan to replace missing items: if one item was missing, the score was not computed.
Time Frame: Baseline (Day 0), Day 60, and Day 180
Population: Only participants with non-missing data at each timepoint were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 97 | 52 | 62 | 28
Score on a scale
  Baseline: number analyzed (Participants) | 21 | 13 | 16 | 7
  Baseline | 21.4 (12.0) | 21.6 (9.4) | 26.6 (14.4) | 19.0 (7.9)
  Day 60: number analyzed (Participants) | 21 | 13 | 14 | 5
  Day 60 | 17.4 (10.7) | 21.3 (9.7) | 27.1 (16.2) | 18.8 (13.8)
  Day 180: number analyzed (Participants) | 17 | 8 | 14 | 6
  Day 180 | 15.4 (11.3) | 24.4 (6.2) | 28.9 (17.0) | 14.8 (11.4)

40. Secondary Outcome: Change From Baseline in the Hypoglycemia Fear Survey, Part 2 (HFS2) Worry Subscale Score at Day 60 and Day 180
Description: as for outcome 39
Time Frame: Baseline (Day 0), Day 60, and Day 180
Population: Only participants with non-missing data at Baseline and Day 60 or Day 180 were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 21 | 13 | 14 | 5
Score on a scale
  Change from Baseline at Day 60 | -4.0 (8.7) | -0.3 (6.8) | -1.4 (7.2) | -1.4 (6.2)
  Change from Baseline at Day 180: number analyzed (Participants) | 17 | 8 | 14 | 5
  Change from Baseline at Day 180 | -5.2 (9.8) | 1.4 (12.5) | 0.9 (10.1) | -3.0 (4.8)

41. Secondary Outcome: Change From Baseline in the Partner Diabetes Distress Scale (Partner-DDS) Questionnaire Total and Subscale Scores at Day 60 and Day 180
Description: The Partner-DDS is a 21-item self-report scale that highlights four critical dimensions of partner-related distress: "my partner's diabetes management", "how best to help", "diabetes and me", and "hypoglycemia". The scale ranges from 0 (not at all) to 4 (a great deal). The Partner-DDS yields a total diabetes distress score plus 4 subscale scores: Total Partner-DDS Score = Mean of the 21 items; My partner's diabetes management = Mean of item 3, 4, 10, 12, 14, 15 and 20; How best to help = Mean of item 2, 6, 7, 11 and 13; Diabetes and me = Mean of items 5, 8, 9, 16 and 21; Hypoglycemia = Mean of items 1, 17, 18 and 19. A lower Partner-DDS score (or a negative change from baseline score) indicates a lower level of distress.
Time Frame: Baseline (Day 0), Day 60, and Day 180
Population: This analysis includes partners with non-missing data (i.e., who filled out the Partner-DDS) for each dimension. The total number of participants analyzed includes the overall number of partners of the participants who had filled out the DDS2 questionnaire.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control - Usual Glucose Monitoring System (SMBG or FGM)
Number analyzed (Participants) | 22 | 14 | 18 | 8
Score on a scale
  My Partner's Diabetes Management - Change from Baseline (BL) at Day 60: number analyzed (Participants) | 2 | 2 | 2 | 2
  My Partner's Diabetes Management - Change from Baseline (BL) at Day 60 | 0.0 (0.4) | 0.1 (0.7) | 0.1 (0.3) | -0.4 (0.4)
  My Partner's Diabetes Management - Change from BL at Day 180: number analyzed (Participants) | 2 | 1 | 2 | 2
  My Partner's Diabetes Management - Change from BL at Day 180 | -1.1 (1.5) | 0.6 (NA) — Standard deviation could not be calculated using data from a single participant. | -0.3 (0.0) | -0.7 (0.2)
  How Best to Help - Change from BL at Day 60: number analyzed (Participants) | 2 | 2 | 2 | 2
  How Best to Help - Change from BL at Day 60 | -1.7 (1.0) | 0.9 (0.1) | 0.1 (0.4) | -0.2 (0.0)
  How Best to Help - Change from BL at Day 180: number analyzed (Participants) | 2 | 1 | 2 | 2
  How Best to Help - Change from BL at Day 180 | -0.5 (0.4) | 1.4 (NA) — Standard deviation could not be calculated using data from a single participant. | -0.8 (0.3) | -0.3 (0.1)
  Diabetes and Me - Change from BL at Day 60: number analyzed (Participants) | 2 | 2 | 2 | 2
  Diabetes and Me - Change from BL at Day 60 | -0.3 (0.7) | 0.2 (0.3) | 0.1 (0.4) | -0.3 (0.4)
  Diabetes and Me - Change from BL at Day 180: number analyzed (Participants) | 2 | 1 | 2 | 2
  Diabetes and Me - Change from BL at Day 180 | 0.3 (0.4) | 0.4 (NA) — Standard deviation could not be calculated using data from a single participant. | -0.9 (0.1) | -0.5 (0.4)
  Hypoglycemia - Change from BL at Day 60: number analyzed (Participants) | 2 | 2 | 2 | 2
  Hypoglycemia - Change from BL at Day 60 | -0.3 (0.0) | -0.1 (0.5) | 0.1 (0.2) | 0.5 (1.1)
  Hypoglycemia - Change from BL at Day 180: number analyzed (Participants) | 2 | 1 | 2 | 2
  Hypoglycemia - Change from BL at Day 180 | 0.6 (1.2) | 0.0 (NA) — Standard deviation could not be calculated using data from a single participant. | 0.4 (0.9) | -0.3 (0.4)
  PDDS Score - Change from BL at Day 60: number analyzed (Participants) | 2 | 2 | 2 | 2
  PDDS Score - Change from BL at Day 60 | -0.5 (0.3) | 0.3 (0.1) | 0.1 (0.3) | -0.2 (0.2)
  PDDS Score - Change from BL at Day 180: number analyzed (Participants) | 2 | 1 | 2 | 2
  PDDS Score - Change from BL at Day 180 | -0.3 (0.9) | 0.6 (NA) — Standard deviation could not be calculated using data from a single participant. | -0.4 (0.2) | -0.5 (0.1)

ADVERSE EVENTS:
Time Frame: From Day 0 (sensor insertion) until Day 180; for Cohort 2, Contol: From Day 0 to Day 120 and From Day 120 to Day 180
Arm/Group | Cohort 1, Enabled - Eversense XL CGM System | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Enabled - Eversense XL CGM System | Cohort 2, Control (Day 0 to 120) - Usual Glucose Monitoring System (SMBG or FGM) | Cohort 2, Control (Day 120 to 180) - Eversense XL CGM System or Usual Glucose Monitoring System
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/52 | 0/62 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 7/97 | 5/52 | 2/62 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 2/97 | 1/52 | 4/62 | 1/28 | 1/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Enabled - Eversense XL CGM System (N=97) | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) (N=52) | Cohort 2, Enabled - Eversense XL CGM System (N=62) | Cohort 2, Control (Day 0 to 120) - Usual Glucose Monitoring System (SMBG or FGM) (N=28) | Cohort 2, Control (Day 120 to 180) - Eversense XL CGM System or Usual Glucose Monitoring System (N=28)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Diabetic ketosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Neuritis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Optic neuritis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Retinopathy proliferative (Eye disorders) | 1 | 0 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Burnout syndrome (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Enabled - Eversense XL CGM System (N=97) | Cohort 1, Control - Usual Glucose Monitoring System (SMBG or FGM) (N=52) | Cohort 2, Enabled - Eversense XL CGM System (N=62) | Cohort 2, Control (Day 0 to 120) - Usual Glucose Monitoring System (SMBG or FGM) (N=28) | Cohort 2, Control (Day 120 to 180) - Eversense XL CGM System or Usual Glucose Monitoring System (N=28)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 4 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT03445065/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT03445065/SAP_001.pdf